CLINICAL TRIAL: NCT00514254
Title: Endometrial Cancer in Black Women
Brief Title: Risk Factors for Endometrial Cancer in Black Women
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); The City College of New York (Other); DOWNSTATE MED/KINGS CO/BKLYN (Unknown); Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 07-093; P30CA008748 (NIH); MSKCC-07093
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; risk factors; questionnaire; 07-093
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva/buccal specimens

GROUPS / COHORTS (2):
- case: Participants complete questionnaires about lifestyle factors and their usual diet and measure their waist and hips. Saliva or buccal specimens are collected for future research.
  Interventions: Other: questionnaire administration; Other: study of socioeconomic and demographic variables; Procedure: evaluation of cancer risk factors
- control: Participants complete questionnaires about lifestyle factors and their usual diet and measure their waist and hips. Saliva or buccal specimens are collected for future research.
  Interventions: Other: questionnaire administration; Other: study of socioeconomic and demographic variables; Procedure: evaluation of cancer risk factors

INTERVENTIONS:
Other: questionnaire administration
Other: study of socioeconomic and demographic variables
Procedure: evaluation of cancer risk factors

SUMMARY:
RATIONALE: Learning about the risk factors for endometrial cancer in black women may help the study of endometrial cancer in the future.

PURPOSE: This clinical trial is studying risk factors for endometrial cancer in black women.

DETAILED DESCRIPTION:
OBJECTIVES:

* Establish and evaluate procedures for conducting a hospital-based case-control study of risk factors for endometrial cancer in black women.

OUTLINE: This is a multicenter study.

Participants complete questionnaires about lifestyle factors and their usual diet and measure their waist and hips. Saliva or buccal specimens are collected for future research.

PROJECTED ACCRUAL:

* A total of 30 cases and 30 controls will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cases

  * Diagnosed with endometrial cancer within the past year
  * Self-identified as being black, African-American, black Hispanic, African, or Afro-Caribbean
* Healthy controls

  * Self-identified as being black, African-American, black Hispanic, African, or Afro-Caribbean
  * No history of endometrial or other cancer (except non-melanoma skin cancer)
  * No prior hysterectomy

PATIENT CHARACTERISTICS:

* Speak English
* No medical condition that would make it difficult to complete the interview

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Black women (including African-American, African, Afro-Caribbean women) with endometrial cancer and controls will be recruited at MSKCC, SUNY Downstate Medical Center and Montefiore Medical Center hospitals. Controls will be black (including African-American, African, Afro-Caribbean) women without history of cancer, who have intact uteri, and will be identified in gynecology clinics. Controls will also be recruited at the Breast Examination Center of Harlem (BECH), an affiliate of MSKCC, providing high quality screening services to a minority community.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2007-07; Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of potential cases and controls approached who are found to be eligible for the study and reasons for being ineligible (including language) | 2 years
Number and percentage of cases and controls approached who sign informed consent | 2 years
Number and percentage of cases and controls who complete each part of the study (main questionnaire, diet questionnaire, saliva/buccal specimen) | 2 years
Proportion of questions with missing data | 2 years
Interviewer's evaluation of interview quality and respondent cooperation | 2 years
Number and percentage of cases who are willing to have tumor specimens used for future research | 2 years
Characteristics of cases and controls (demographics, main risk factors, and use of health care and screening) | 2 years
Proportion of participants who rate the study positively on each measure in the post-interview assessment and respondents' suggested changes to the study | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sara Olson, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - SUNY Downstate Medical Center, Brooklyn, New York
  - City College of New York, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm